CLINICAL TRIAL: NCT00721266
Title: An Open Label, Dose-escalation Study to Evaluate Safety, Pharmacokinetics and Tumor Growth Control Rate of RO5083945, a Glycoengineered Antibody Against EGFR, in Patients With Metastatic and/or Locally Advanced Malignant EGFR+ Solid Tumors.
Brief Title: A Dose-Escalation Study of RO5083945 in Patients With Metastatic and/or Locally Advanced Malignant Epidermal Growth Factor Receptor (EGFR)+ Solid Tumors.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BO21495; 2007-005939-28
Record Dates: First submitted 2008-07-04; First posted 2008-07-24 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — imgatuzumab

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: RO5083945

INTERVENTIONS:
Drug: RO5083945 — Administered iv, either weekly, every 2 weeks or every 3 weeks, at escalating doses (with a starting dose of 50mg weekly (Part 1)). Recommended dose administered iv, either weekly, every 2 weeks or every 3 weeks (Part 2).

SUMMARY:
This study will evaluate the pharmacokinetics, maximum tolerated dose and anti-tumor activity of RO5083945 in patients with metastatic and/or locally advanced malignant EGFR+ solid tumors. In the first part of the study, groups of patients will be sequentially enrolled to receive ascending doses of RO5083945 administered weekly, every 2 weeks or every 3 weeks. The starting dose of 50mg weekly will be escalated in subsequent groups of patients after a successful assessment of the safety, tolerability and pharmacokinetics of the previous dose. In Part 2 of the study, patients with EGFR+ and mutant KRAS colorectal cancer will be enrolled, and will receive RO5083945 at the recommended dose and regimen identified in Part 1. The anticipated time on study treatment is until disease progression, and the target sample size is <100 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >=18 years of age;
* centrally confirmed EGFR expression in tumor tissue;
* radiologically measurable or clinically evaluable disease;
* last dose of systemic anti-neoplastic therapy or radiotherapy >=28 days prior to start of study;
* histologically or cytologically confirmed advanced stage, primary or metastatic EGFR+ solid tumors (Part 1);
* histologically or cytologically confirmed advanced stage, primary or metastatic EGFR+ and mutant KRAS colorectal cancer (Part 2);
* not more than 2 previous cytotoxic regimens for metastatic disease (Part 2).

Exclusion Criteria:

* history of grade 3-4 toxicity resulting from previous anti-EGFR treatment;
* known or suspected CNS metastases;
* wild type KRAS colorectal cancer (Part 2).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2008-06; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameters, and maximum tolerated dose (Part 1) | Throughout study
Tumor growth control rate (CR, PR, SD) (Part 2) | Event driven

SECONDARY OUTCOMES:
AEs and laboratory parameters, pharmacodynamic parameters (Parts 1 and 2) | Throughout study
Anti-tumor activity (ORR, DR, PFS) (Part 2) | Event driven

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (5):
- France (2):
  - Toulouse
  - Villejuif
- Spain (3):
  - Barcelona, Barcelona
  - Seville, Sevilla
  - Valencia, Valencia

REFERENCES:
- [Derived] Paz-Ares LG, Gomez-Roca C, Delord JP, Cervantes A, Markman B, Corral J, Soria JC, Berge Y, Roda D, Russell-Yarde F, Hollingsworth S, Baselga J, Umana P, Manenti L, Tabernero J. Phase I pharmacokinetic and pharmacodynamic dose-escalation study of RG7160 (GA201), the first glycoengineered monoclonal antibody against the epidermal growth factor receptor, in patients with advanced solid tumors. J Clin Oncol. 2011 Oct 1;29(28):3783-90. doi: 10.1200/JCO.2011.34.8888. Epub 2011 Sep 6. PMID 21900113